CLINICAL TRIAL: NCT04950348
Title: Preliminary Exploration of Clinical Trials of Prosthesis and Surgery Guide System for Personalized Total Knee Arthroplasty
Brief Title: Clinical Trials of Prosthesis and Surgery Guide System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Inner Mongolia People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M2020519
Record Dates: First submitted 2021-06-25; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printed personalized TKA prosthesis (Experimental): Patients in the experimental group received 3D printed personalized TKA prosthesis treatment
  Interventions: Device: Personalized TKA prosthesis
- Zimmer NexGen TKA prostheses (Active Comparator): Patients in the active comparator group received Zimmer NexGen TKA prostheses treatment
  Interventions: Device: Zimmer NexGen prostheses

INTERVENTIONS:
Device: Personalized TKA prosthesis — TKA prosthesis that is designed and manufactured according to the patient's knee joint anatomy
  Arms: 3D printed personalized TKA prosthesis
Device: Zimmer NexGen prostheses — Commercial products used on a large scale
  Arms: Zimmer NexGen TKA prostheses

SUMMARY:
1. The subject continues the research of Professor JiaKuo Yu's research group on the personalized design, processing and manufacturing of personalized total knee replacement artificial joint prostheses and the verification of animal and human cadavers. It is planned to carry out the femoral condyle prosthesis of personalized total knee replacement prosthesis. Clinical trials are carried out on the body, tibial tray prosthesis and meniscus prosthesis; at the same time, in order to achieve personalized precision surgery, the clinical trial verification is carried out on the placement of personalized surgical guides that match the personalized artificial joints.
2. In the clinical verification study, the research team will summarize the role of personalized artificial joints for total knee replacement and personalized implant surgical guides in the precise and minimally invasive treatment of knee joint diseases.

DETAILED DESCRIPTION:
This study aims to evaluate the safety and effectiveness of the femoral condyle prosthesis, tibial tray prosthesis and meniscus prosthesis of the personalized total knee replacement system; to verify the clinical feasibility and safety of the personalized surgical guide, as a personalized total knee replacement The clinical application of the prosthesis and its guide lays the foundation, including:

2.1 Evaluate the advantages of personalized total knee replacement surgery in osteotomy methods, evaluate the impact of anatomical osteotomy methods on intraoperative and postoperative effects and early and long-term clinical effects.

2.2 By measuring the amount of osteotomy in personalized total knee replacement surgery, evaluate the impact of a smaller and reasonable amount of osteotomy on the patient's early and long-term clinical results.

2.3 Verify the clinical effect of personalized total knee replacement prosthesis, and provide the basis for its clinical promotion and application.

ELIGIBILITY:
Inclusion Criteria:

1. Degenerative osteoarthritis, traumatic arthritis or avascular necrosis, inflammatory joint disease and other end-stage knee joint diseases, as well as the correction of deformities, reconstruction after failure of some knee joint prostheses, and other techniques that cannot be handled In the case of fractures, total knee prosthesis replacement is required.
2. Age ≥50, ≤80 years old.
3. The subject or guardian is willing and able to sign an informed consent form.

Exclusion Criteria:

1. History of previous knee surgery.
2. Severe knee joint deformity (valgus greater than 15° or valgus greater than 20°) or knee joint instability;
3. Severe flexion contracture deformity (flexion contracture> 25°);
4. Perform total knee joint revision and replacement surgery;
5. Rheumatoid arthritis;
6. Body mass index (BMI)> 35.;
7. Patients with neuromuscular insufficiency (for example: paralysis, myolysis or muscle weakness) can lead to postoperative knee instability or abnormal gait;
8. Pregnant or lactating women;
9. Suffer from the underlying medical condition (including but not limited to metabolism, hematology, kidney, liver, lung, nerve, endocrine, heart, infection or gastrointestinal tract) that the researcher believes that the patient is at an unacceptable risk; Serious progressive or uncontrolled diseases that are not suitable for trials or put them at high risk, including any medical or psychiatric conditions that the investigator believes will prevent the subject from following the protocol or completing the study according to the protocol;
10. Being infected with human immunodeficiency virus (HIV), infectious hepatitis B or hepatitis C or corresponding medical history;
11. Suffering from a progressive infection or malignant disease, can provide chest X-ray, computed tomography (CT scan) or MRI evidence within 12 weeks before screening, and it is verified by a qualified physician.
12. Active systemic infections (except colds) or any other infections that will recur regularly during the previous two weeks;
13. There is a history of chronic or recurrent infectious diseases, or evidence of tuberculosis infection that was determined to be positive at the time of screening. Subjects who have obtained positive or uncertain results can participate in the study if they have undergone a comprehensive tuberculosis examination (according to local practice/guidelines) within 12 weeks before baseline and finally confirmed that there is no evidence of active tuberculosis. If the presence of latent tuberculosis is confirmed, treatment must be initiated and maintained in accordance with local or national guidelines before the baseline;
14. History of lymphoproliferative disease, or any known malignant tumor, or history of malignant tumor of any organ system in the past 5 years (Bowen's disease, basal cell carcinoma, or actinic keratosis after treatment and no evidence of recurrence in the past 12 weeks Except for diseases; except for excised cervical carcinoma in situ or non-invasive malignant colon polyps);
15. Suffer from medical problems at the same time, including but not limited to the following:

(1) Uncontrolled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥95mmHg), congestive heart failure (New York Heart Association status classification III or IV); (2) Subjects whose serum creatinine level exceeds 2.0 mg/dl (176.8 μmol/L); (3) Total white blood cell (WBC) count at screening <2500/μL, or platelet <100000/μL or neutrophil <1500/μL or hemoglobin <8.5 g/dL; (4) Within six months before the baseline, there is a history of alcohol or drug abuse or evidence of ongoing abuse.

16) The patient is mentally incapable or unable to understand the requirements for participating in the research.

Ages: 51 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Mechanical axis of the lower limb and prosthesis position | 7 days postoperatively
  Axis through the center of the hip joint, the center of the knee joint, and the center, (-3,3) is normal.
Mechanical axis of the lower limb and prosthesis position | 3months postoperatively
  Axis through the center of the hip joint, the center of the knee joint, and the center, (-3,3) is normal.
Mechanical axis of the lower limb and prosthesis position | 6 months postoperatively
  Axis through the center of the hip joint, the center of the knee joint, and the center, (-3,3) is normal.
Mechanical axis of the lower limb and prosthesis position | 12 months postoperatively
  Axis through the center of the hip joint, the center of the knee joint, and the center, (-3,3) is normal.

SECONDARY OUTCOMES:
Osteotomy | during surgery
  The size of the osteotomy
Operation time | during surgery
  Operation time

OTHER OUTCOMES:
KSS score | 7 days，3months， 6 months and 12 months postoperatively
  knee society score, the scale is 0-200 and 0 is worse.
WOMAC score | 7 days，3months， 6 months and 12 months postoperatively
  The Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index, the scale is 0-100 and 100 is worse.
SF-36 score | 7 days，3months， 6 months and 12 months postoperatively
  short form 36 questionnaire, scale is 0-100 and 0 is worse.

CONTACTS AND LOCATIONS:
Overall Officials: Jia-kuo Yu, Prof., Study Chair — Peking University Third Hospital
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No